CLINICAL TRIAL: NCT02424032
Title: Stabilization Exercises With and Without Connective Tissue Massage for Chronic Mechanical Neck Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seyda TOPRAK CELENAY (Other)
Responsible Party: Sponsor-Investigator, Seyda TOPRAK CELENAY, Assistant Professor, Ataturk Training and Research Hospital
Organization: Ataturk Training and Research Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: GO 13/381
Record Dates: First submitted 2015-04-08; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Neck Pain Musculoskeletal
Keywords: Neck pain; stabilization exercise; connective tissue massage
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Exercise and connective tissue massage (Experimental): Stabilization exercise and connective tissue massage have been applied
  Interventions: Behavioral: "Exercise" and "connective tissue massage"
- Exercise (Active Comparator): Only stabilization exercise has been applied
  Interventions: Behavioral: "Exercise"

INTERVENTIONS:
Behavioral: "Exercise" and "connective tissue massage" — Cervical and scapulothoracic stabilization exercises with connective tissue massage were performed.The program was carried out for 12 sessions, 3 days/week in 4 weeks.
  Arms: Exercise and connective tissue massage
Behavioral: "Exercise" — Cervical and scapulothoracic stabilization exercises were performed. The program was carried out for 12 sessions, 3 days/week in 4 weeks.
  Arms: Exercise

SUMMARY:
The aim of this study was to investigate and compared the effects of cervical and scapulothoracic stabilization exercises with and without connective tissue massage (CTM) for patients with chronic mechanical neck pain.

DETAILED DESCRIPTION:
Sixty patients with chronic mechanical neck pain were recruited and randomly allocated into stabilization exercise with and without the connective tissue massage program. The study's inclusion criteria were as follows: 18 to 65 years of age, having neck pain for more than 3 months, and being volunteer. The exclusion criteria were as follows: stenosis, traumatic injury history, previous surgery related to cervical spine, hypermobility, cancer, having inflammatory rheumatologic, severe psychological disorders, being pregnant, and intervention including exercise or physical therapy in the last 3 months.The program was carried out for 12 sessions, 3 days/week in 4 weeks. Pain intensity with Visual Analog Scale, pressure pain threshold with digital algometer, the level of anxiety with the Spielberger State Trait Anxiety Inventory, and life quality with Short Form-36 were evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age,
* having neck pain for more than 3 months, and
* being volunteer

Exclusion Criteria:

* Stenosis,
* traumatic injury history,
* previous surgery related to cervical spine,
* hypermobility,
* cancer,
* having inflammatory rheumatologic,
* severe psychological disorders,
* being pregnant, and
* intervention including exercise or physical therapy in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Change in Neck pain intensity as measured by Visual Analog Scale | Change from baseline neck pain intensity at 4 weeks

SECONDARY OUTCOMES:
Change in level of anxiety as assessed by Spielberger State Trait Anxiety Inventory | Change from baseline level of anxiety at 4 weeks
Change in quality of life as assessed by Short Form-36 | Change from baseline quality of life at 4 weeks
Change in pressure pain threshold as measured by digital algometer | Change from baseline pressure pain threshold at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seyda TOPRAK CELENAY, Principal Investigator — Ataturk Trainning and Research Hospital
Locations (1):
- Ataturk Trainning and Research Hospital, Ankara, Cankaya, Turkey (Türkiye)

REFERENCES:
- [Result] Bakar Y, Sertel M, Ozturk A, Yumin ET, Tatarli N, Ankarali H. Short term effects of classic massage compared to connective tissue massage on pressure pain threshold and muscle relaxation response in women with chronic neck pain: a preliminary study. J Manipulative Physiol Ther. 2014 Jul-Aug;37(6):415-21. doi: 10.1016/j.jmpt.2014.05.004. Epub 2014 Aug 6. PMID 25108749
- [Result] Dusunceli Y, Ozturk C, Atamaz F, Hepguler S, Durmaz B. Efficacy of neck stabilization exercises for neck pain: a randomized controlled study. J Rehabil Med. 2009 Jul;41(8):626-31. doi: 10.2340/16501977-0392. PMID 19565156
- [Result] Jull G, Trott P, Potter H, Zito G, Niere K, Shirley D, Emberson J, Marschner I, Richardson C. A randomized controlled trial of exercise and manipulative therapy for cervicogenic headache. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1835-43; discussion 1843. doi: 10.1097/00007632-200209010-00004. PMID 12221344
- [Result] Sherman KJ, Cherkin DC, Hawkes RJ, Miglioretti DL, Deyo RA. Randomized trial of therapeutic massage for chronic neck pain. Clin J Pain. 2009 Mar-Apr;25(3):233-8. doi: 10.1097/AJP.0b013e31818b7912. PMID 19333174
- [Derived] Celenay ST, Kaya DO, Akbayrak T. Cervical and scapulothoracic stabilization exercises with and without connective tissue massage for chronic mechanical neck pain: A prospective, randomised controlled trial. Man Ther. 2016 Feb;21:144-50. doi: 10.1016/j.math.2015.07.003. Epub 2015 Jul 15. PMID 26211422